CLINICAL TRIAL: NCT06302478
Title: Effects of a Venous Thromboembolism Prevention Program on the Occurrence of Venous Thromboembolism in Patients With Spinal Cord Disorders
Brief Title: 5E Program for Preventing Venous Thromboembolism in Patients With Spinal Cord Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Wiphawadee Potisopha, Principle Investigator, Khon Kaen University
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: KhonKaenU001
Record Dates: First submitted 2024-01-21; First posted 2024-03-08 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Venous Thromboembolism; Spinal Cord Diseases; Spinal Cord Injuries; Nurse's Role
MeSH Terms: conditions — Venous Thromboembolism; Spinal Cord Diseases; Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: A quasi-experimental research (two group pretest-posttest design)
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5E Program (Experimental): Participants in the 5E program group will receive 7-day nursing interventions.
  Interventions: Behavioral: 5E program
- Usual Care (No Intervention): Participants in the control group will receive 7-day usual care interventions, including health education regarding signs and symptoms of venous thromboembolism and IPC use if the participants experienced muscle power as grade 0.

INTERVENTIONS:
Behavioral: 5E program — Participants in the 5E program group will receive 7-day nursing interventions including
  * Education: health education regarding venous thromboembolism prevention
  * Elevation: leg elevation of 10-20 degrees
  * Exercise: ankle exercises
  * Enough fluid: adequate fluid uptake
  * Early application of intermittent pneumatic compression (IPC): IPC use within 48 hours after admission
  Arms: 5E Program

SUMMARY:
The goal of this quasi-experimental study is to examine the effects of a venous thromboembolism prevention program, or "5E" program, on the rates of venous thromboembolism in patients with spinal cord disorders. The main questions it aims to answer are:

* Will participants receiving the 5E program have lower rates of venous thromboembolism compared to those receiving the usual care?
* Will participants receiving the 5E program have lower scores of venous thromboembolism signs and symptoms compared to those receiving the usual care?
* Will the average thigh and calf circumferences of participants before and after receiving the 5E program be different?

Participants in the intervention group will receive the 5E program, including

* Education: health education regarding venous thromboembolism prevention
* Elevation: leg elevation of 10-20 degrees
* Exercise: ankle exercises
* Enough fluid: adequate fluid uptake
* Early application of intermittent pneumatic compression (IPC): IPC use within 48 hours after admission

ELIGIBILITY:
Inclusion Criteria:

* Caprini scores of 5-8 and >8
* Able to communicate in the Thai language
* Willing to participate in this study

Exclusion Criteria:

* Alteration of consciousness
* Experiencing complications, including neurogenic shock and autonomic dysreflexia
* Being pregnant
* Having fluid restriction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
The rate of venous thromboembolism | The day before implementing the intervention and at 7 days after implementing intervention
  The diagnosis of venous thromboembolism is confirmed by a Doppler ultrasound scan of the femoral vein and popliteal vein by a physician working at the study site. The physician will record the results in the data record form.

SECONDARY OUTCOMES:
Signs and symptoms of deep venous thrombosis and pulmonary embolism | The day before implementing the intervention and Day 1 - Day 7 after implementing intervention
  The Well's Score for deep venous thrombosis (DVT) includes clinical parameters: active cancer or palliative (+1), paralysis (+1), recently bedridden for more than 3 days (+1), localized tenderness (+1), entire leg swelling (+1), calf swelling more than 3 cm compared with asymptomatic leg (+1), pitting edema (+1), previous DVT documented (+1), collateral superficial veins (non-varicose) (+1), and alternative diagnosis (-2).
  The Modified Well's Score for pulmonary embolism (PE) includes the following criteria: clinical signs and symptoms of DVT (3); an alternative diagnosis is less likely than PE (3); a heart rate greater than 100 (1.5); immobilization for 3 or more consecutive days (1.5); previous objectively diagnosed PE or DVT (1.5); hemoptysis (1); and malignancy (1).
Thigh and calf circumference | The day before implementing the intervention and Day 1 - Day 7 after implementing intervention
  Thigh and calf circumferences will be measured in centimeters using the standardized measuring tape. The assistant researcher will record the results in the data record form.

CONTACTS AND LOCATIONS:
Locations (1):
- Chaiyaphum Hospital, Chaiyaphum, Thailand